CLINICAL TRIAL: NCT07097545
Title: Social Media Use Study
Brief Title: Change in Social Media Use and Well-being Among College Students Receiving a Two-week Exercise or Mindfulness Intervention
Acronym: SMUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00025926-RCT2
Record Dates: First submitted 2025-07-25; First posted 2025-07-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Social Media Addiction; Anxiety; Depression Disorder; Wellbeing
Keywords: digital media reduction intervention; mindfulness; behavioral intervention; digital wellbeing
MeSH Terms: conditions — Internet Addiction Disorder; Anxiety Disorders | interventions — Mindfulness; Exercise

STUDY DESIGN:
Intervention Model Description: Three groups of 1) no intervention, 2) mindfulness, or 3) social media reduction + exercise replacement intervention arms
Masking Description: Both participants and investigators will know which intervention group each participant has been randomized into.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants will not receive an intervention. Participants will receive instructions to use social media use as usual.
- Mindfulness (Experimental): Approximately 15 minute mindfulness style meditations will be completed daily for two weeks through the Calm platform. Participants can listen to the exercise on the web-enabled version of Calm, or through the smartphone app. The first course is entitled "7 Days of Gratitude" and centers around noticing and appreciating things in daily life, the second course is entitled "7 Days of managing stress" that focuses on building awareness and coping with that specific area of mental stress, such as de-escalating stress, mind-body connection, strong emotions, negative self-talk, and how events are interpreted.
  Interventions: Behavioral: Mindfulness
- Social Media Reduction + Exercise (Experimental): Participants will reduce social media use by at least 30 minutes daily for two weeks. Simultaneously, participants will exercise at least 30 minutes daily. Participants are given examples of common exercises (walking, yoga, strength training, etc.), but are allowed to choose any type, although dissuaded from activities with high potential for injury.
  Interventions: Behavioral: Social Media Reduction; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Mindfulness — 15 minute daily guided meditation
  Arms: Mindfulness
Behavioral: Social Media Reduction — Reduce social media use at least 30 minutes daily and exercise instead
  Arms: Social Media Reduction + Exercise
Behavioral: Exercise — Participants will exercise at least 30 minutes daily. Participants are given examples of common exercises (walking, yoga, strength training, etc.), but are allowed to choose any type, although dissuaded from activities with high potential for injury.
  Arms: Social Media Reduction + Exercise

SUMMARY:
The investigators will be randomizing 300 college student participants with high levels of social media use into either a 1) control condition (no intervention), a 2) mindfulness meditation cognitive intervention, or 3) a social media reduction + exercise replacement intervention. Participants complete intervention activities daily for two weeks. The investigators will collect self-report and behavioral measures of social media use and related psychological constructs at three time points: baseline, immediately after the intervention period, and one-week after the intervention period (three weeks from baseline).

DETAILED DESCRIPTION:
The objective of this study is to test two cognitive and behavioral interventions designed to reduce social media use and improve psychological constructs related to social media use in a sample of university students. The cognitive intervention is a mindfulness meditation exercise taken from the Calm app focused around gratitude and stress management. Each meditation takes approximately 15 minutes to complete and is to be done daily for two week. The second behavioral intervention is asking participants to reduce social media use for 30 minutes daily for two weeks and replacing that time with physical exercise of the participants' choosing.

Aim 1: Compare psychological constructs related to mental health (well-being, stress, depression, anxiety, loneliness, social comparisons, etc.) before and after conducting two social media use interventions over two weeks, compared to a control condition (no intervention).

Aim 2: Compare self-reported and behavioral (smartphone screenshots of social media use screentime) measures of social media use before and after two social media use interventions over two weeks, compared to a control condition (no intervention).

Aim 3: Examine mental health and social media use one week after the intervention period is complete (3-week follow up) or testing whether the interventions have effects beyond the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* The participant is 18 or older.
* The participant must be a Johns Hopkins University student.
* Owning an iPhone or Android smartphone, with frequent use of social media use daily (>

  1 hour)
* Enabling and sharing screenshots of the participant's smartphone use metrics, including number of last-week pickups, notifications received, and average screen time.
* Providing consent to participate.
* Only exercising 1 hour or less daily, on average.

Exclusion Criteria:

* younger than 18
* Not a Johns Hopkins University Student
* Doesn't own a smart phone
* Uses smartphone less than 1 hour daily
* Exercises more than 1 hour daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Depression, Anxiety and Stress Scale - 21 (DASS-21) | baseline, immediately post intervention, post intervention up to one week
  Score range = 0-63, higher score = worse outcome
Change in World Health Organization Quality of Life (WHOQoLBREF) scale | baseline, immediately post intervention, post intervention up to one week
  Score range = 13-65, lower score = worse outcome
Change in smartphone screen time (minutes) for social media use | baseline, immediately post intervention, post intervention up to one week
  Past-week amount of screen time for social media use
Change in number of social media use smartphone pick-ups | baseline, immediately post intervention, post intervention up to one week
  Past-week total number of smartphone pickups for social media use applications
Change in percent of time using social media | baseline, immediately post intervention, post intervention up to one week
  Past-week percent of time using social media compared to other smartphone application categories.
Change in social media use notifications received | baseline, immediately post intervention, post intervention up to one week
  Past-week total number of notifications received for social media use applications

SECONDARY OUTCOMES:
Change in University of California, Los Angeles 3-Item Loneliness Scale | baseline, immediately post intervention, post intervention up to one week
  Score range = 3-9, higher score = worse outcome
Change in The Gratitude Questionnaire, 6-item form (GQ-6) scale | baseline, immediately post intervention, post intervention up to one week
  Score range = 6-42, lower score = worse outcome
Change in Motivations for Electronic Interaction Scale (MEIS) | baseline, immediately post intervention, post intervention up to one week
  Score range = 10-50, higher score = worse outcome
Change in Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT-15) | baseline, immediately post intervention, post intervention up to one week
  scale Score range = 0-138, lower scores = worse outcome
Change in Bergen Social Media Addiction Scale (BSMAS) | baseline, immediately post intervention, post intervention up to one week
  Score range = 6-35, higher score = worse outcome
Change in Fear of Missing Out Scale | baseline, immediately post intervention, post intervention up to one week
  Score range = 10-50, higher score = worse outcome
Change in hours spent socializing inperson with peers | baseline, immediately post intervention, post intervention up to one week
  Score range = 0-20+ hours of in-person socialization, lower scores = worse outcome
Change in number of evenings of past-week recreation | baseline, immediately post intervention, post intervention up to one week
  Score range = 0-7 evenings of recreation, lower scores = worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Thrul, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and other resources will be shared upon reasonable request.